CLINICAL TRIAL: NCT05375487
Title: The Effect of Natural Carbonated Mineral Water Consumption on Gastrointestinal Transit and on Gut Microbiota in Subjects With Functional Constipation: A Randomized, Placebo-Controlled Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: CINTESIS - Center for Health Technology and Services Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MineralWaterGut
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Functional Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbonated Natural Mineral Water (Experimental): 750 mL/day of carbonated natural mineral water, with high content of bicarbonate, calcium and magnesium.
  Interventions: Other: Carbonated Natural Mineral Water
- Low Mineral Water (Placebo Comparator): 750 mL/day of low mineral water.
  Interventions: Other: Low Mineral Water

INTERVENTIONS:
Other: Carbonated Natural Mineral Water — 750 mL/day of carbonated natural mineral water, with high content of bicarbonate, calcium, and magnesium, in three portions of 250 mL (one portion 30 minutes prior to lunch, one during the afternoon and the last portion minutes before dinner), during 4 weeks.
  Arms: Carbonated Natural Mineral Water
Other: Low Mineral Water — 750 mL/day of low mineral water (one third prior to lunch, one third during the afternoon and the last third 30 minutes before dinner), during 4 weeks.
  Arms: Low Mineral Water

SUMMARY:
Functional constipation (FC) is a common condition associated with aging, lower socioeconomic status, low physical activity and also with reduced fibre, water and magnesium intakes. Different studies have reported a positive association between the intake of hyper-mineral water containing a high content of bicarbonate, calcium, or magnesium, and the improve of the gastrointestinal transit. There is evidence that magnesium and sulphate, both individually, have a laxative action. However, the impact of other minerals is scarce. It has been described different mechanisms explaining how gut microbiota influence the gastrointestinal transit. Specifically, in FC patients, it is important to understand the particularities of their gut microbiota and understand whether the intake of hyper-mineral water, a natural source of minerals, can modify positively the gut microbiota. The aim of the present randomized placebo-controlled pilot trial is to evaluate, for the first time, the effect of the carbonated mineral water consumption in the gastrointestinal transit and in the gut microbiota of subjects with FC.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 70
* Having Functional Constipation diagnosis criteria, according to the Rome IV criteria
* Not using any laxative drug for 3 days before screening visit
* Drinking 1.0 ± 0.5 L of water per day
* Accept and sign the consent

Exclusion Criteria:

* Treatment or disease (current or past) likely to interfere with evaluation of the study parameters
* Taking antibiotics in the 3 months preceding the recruitment visit
* Taking supplements and any food enriched or presented containing bacteria or yeasts likely to have an effect on the gastrointestinal tract, particularly on intestinal transit, digestive comfort, gas production, the occurrence of abdominal pain in the 30 days preceding the recruitment visit (these products will also be banned during the study period)
* Subject having an alcohol consumption of more than 3 glasses of wine a day, or 2 glasses of beer a day, or 1 glass of hard liquor a day
* Subject having a coffee consumption greater than 5 cups per day
* Subject with constipation attributable to an organic or anatomical cause (Hirschsprung's disease, hypothyroidism, mental deficiency, psychiatric illness, neurological abnormalities, history of operation of the colon or anus, colorectal cancer, anemia, etc.)
* Subject with a history of current gastrointestinal pathology or disorder such as duodenal ulcer, chronic colitis, or chronic inflammatory disease of the gastrointestinal tract (Crohn's disease, ulcerative colitis), celiac disease or syndrome irritable bowel
* Subject having a history of operation of the digestive tract
* Subject having undergone surgery in the two months preceding the recruitment visit
* Subject having undergone bariatric surgery
* History of renal disease (renal insufficiency etc.) or cardiovascular disease (cardiac insufficiency...), respiratory disease, neural disease
* Having participated in a weight loss program (with a 5-10% weight) loss in the last 3 months prior to the recruitment visit
* Body mass index > 35 kg/ m2
* Taking supplements of magnesium, vitamins, or other minerals during the study period
* Intake of other carbonated mineral waters beyond the given water, during the study period.
* Pregnancy
* Participation in another clinical trial during the last 30 days prior to the recruitment visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Difference between the intervention and control group in the change in gastrointestinal transit from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in gastrointestinal transit measured by the percentage of responder subjects defined as a composite score of the two following Rome IV criteria: number of stools ≥ 4 or an increase of 2 stools/week and stools consistency with less than 25% of lumpy to hard stools.

SECONDARY OUTCOMES:
Difference between the intervention and control group in the change in stool consistency from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in stool consistency measured using Bristol scale.
Difference between the intervention and control group in the change in constipation symptoms from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in constipation symptoms measured using a validated PAC-SYM questionnaire. PAC-SYM is a 12-item, self-administered questionnaire used to measure severity of symptoms over the past 2 weeks in patients with constipation. Cultural adaptation and linguistic validation of the PAC-SYM for Portugal was performed by Mapi Research.
Difference between the intervention and control group in the change in constipation Quality of Life from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in constipation Quality of Life measured using a validated PAC-QOL questionnaire. PAC-QOL questionnaire is a 28-item self-administered questionnaire that is being used to measure health-related quality of life (over the past 2 weeks) in patients with chronic constipation. Cultural adaptation and linguistic validation of the PAC-QOL for Portugal was performed by Mapi Research Trust.
Difference between the intervention and control group in the change in Perceived Stress Scale from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in constipation Perceived Stress Scale measured using a validated Perceived Stress Scale questionnaire. A validated Perceived Stress Scale (PSS) self-administered questionnaire with 13-item will be used to measure perceived stress of respondents during the last month (Portuguese version keeps 13 of the 14 original items). The PSS questionnaire has been demonstrated to have internal consistency, reproducibility, validity, and sensitivity. Cultural adaptation and linguistic validation of the PSS for Portugal was implemented by Pais-Ribeiro & Marques (2009).
Difference between the intervention and control group in the change in gut microbiota from baseline to the end of follow-up (4 weeks). | 4 weeks
  Bacterial DNA will be extracted from fecal samples. 16SRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Difference between the intervention and control group in the change in short-chain fatty acid profiling from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in short-chain fatty acid profiling evaluated by the faeces concentration of short-chain fatty acids before and after intervention.
Difference between the intervention and control group in the change in urinary excretion of minerals from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in urinary excretion of minerals evaluated by the K+, Na+, Mg2+ and Ca2+ excretion before and after intervention.
Difference between the intervention and control group in the change in urinary pH from baseline to the end of follow-up (4 weeks). | 4 weeks
  Change in urinary pH evaluated by the urine pH before and after intervention.

OTHER OUTCOMES:
Adverse events | 4 weeks
  Registration of any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa; André Rosário, PhD, Study Director — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa; Inês Mota, Study Director — NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA de Lisboa
Locations (1):
- NOVA Medical School | Faculdade de Ciências Médicas da Universidade NOVA, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided